CLINICAL TRIAL: NCT06065332
Title: Randomized Split-Face Study Using a Post-Procedural Biotech Cellulose Mask to Improve Patient Comfort & Downtime
Brief Title: Post-Procedural Biotech Cellulose Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siperstein Dermatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Velez
Record Dates: First submitted 2023-09-20; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The blind evaluator were not aware which side of the face received the mask
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Velez Intense Hydration Mask® (biotech cellulose face mask) Right Side (Experimental): For 30 minutes after an aesthetic procedure, a Velez Intense Hydration Mask® (biotech cellulose face mask) was applied to the right side of the face
  Interventions: Other: Velez Intense Hydration Mask® (biotech cellulose face mask)
- Velez Intense Hydration Mask® (biotech cellulose face mask) Left Side (Experimental): For 30 minutes after an aesthetic procedure, a Velez Intense Hydration Mask® (biotech cellulose face mask) was applied to the left side of the face
  Interventions: Other: Velez Intense Hydration Mask® (biotech cellulose face mask)

INTERVENTIONS:
Other: Velez Intense Hydration Mask® (biotech cellulose face mask) — Application to one randomized side half of a Velez Intense Hydration Mask® (biotech cellulose face mask)

SUMMARY:
Background: There are many post-procedural treatments touted to improve comfort and decrease downtime, but very few prospective randomized studies.

Aims: To analyze the safety and efficacy of a post-procedural biotech cellulose mask Patients/Method: Fifteen patients undergoing either a microneedling with radiofrequency (n=5), non-ablative fractional (n=5), or full erbium;YAG resurfacing (n=5) treatment were randomized to receive a Velez biotech cellulose mask on one side of the face for 30 minutes after the procedure and for two hours a day until healed. Canfield Visia photos and thermal photographs were taken 30 minutes after the procedure and daily until healed. The investigator and blind evaluators reviewed the photos and subjects answered daily questionnaires.

DETAILED DESCRIPTION:
A dual center study was performed at a private practice in Boynton Beach and Boca Raton Florida. The study was carried out in accordance with the ethical guidelines and principles of the 1975 Declaration of Helsinki and good clinical practice. The protocol was approved on May 12th, 2022, by Sterling IRB.

Study Design:

The clinical research coordinator and investigator recruited, enrolled, and assigned 15 subjects into 3 arms, each with 5 subjects over two months. The side assigned a biotech cellulose mask for each subject was determined by random sorting using a computer-generated sequence and written on a label adhered to the mask packaging so the patient could remember while at home.

Treatment:

Topical anesthetic cream (benzocaine 20%, lidocaine 10%, and tetracaine 6%) was applied to the face for 30 minutes and wiped off with 70% isopropyl alcohol in all three arms. Those in arm 1 received a non-ablative fractionated thulium treatment (Moxi; Sciton) those in arm 2 received a microneedling with radiofrequency treatment (Secret; Cutera), and those in arm 3 received a fully ablative erbium yttrium aluminum garnet (Er:YAG) laser resurfacing (Contour TRL; Sciton). Immediately after the procedure a biotech cellulose mask was applied (Hydration mask; Velez by Vesna) and left on for thirty minutes. Then digital photography using Canfield's imaging system and Flir's thermal camera was done. In addition, a subject questionnaire on satisfaction, erythema, edema, and pain levels after the procedure was completed. Patients used the typical post-care treatment on both sides of their face such as Vaseline for laser resurfacing and a hydrating serum for the NAFR and MRF. They were given additional half-sided masks to apply to the same assigned side of their face at home for at least two hours each day for the duration of the study. They returned to the office daily for questionnaires and photographs until deemed fully healed by the primary investigator signifying the end of the study. At all follow up visits, the primary investigator assessed the subject for any side effects and subjects were asked about side effects in questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to undergo a cosmetic procedure
* Patients willing to apply a mask for 30 minutes after the procedure and daily
* Patients willing to return to the office to take photos daily and allow use of photos in publication

Exclusion Criteria:

* History of auto-immune conditions
* History of keloids
* History of severe anaphylactic reactions
* Patients taking either anti-coagulants, chemotherapy, immunosuppressive agents, immunomodulatory agents, diuretics, antihistamines, or anti-inflammatory two weeks before or during planned treatments
* Patients who are pregnant or nursing.

Ages: 22 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Temperature | 30 minutes after the procedure
  Change in skin temperature

CONTACTS AND LOCATIONS:
Overall Officials: Robyn D Siperstein, MD, Principal Investigator — Siperstein Dermatology Group
Locations (1):
- Siperstein Dermatology Group, Boynton Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT06065332/Prot_SAP_000.pdf